CLINICAL TRIAL: NCT07037394
Title: Comparison of Efficacy of Rifaximin, Probiotics and LOLA (L-Ornithine L-Aspartate) in Overt Hepatic Encephalopathy: A Randomized, Phase-IV, Lactulose Controlled Clinical Trial.
Brief Title: A Trial for Comparing Rifaximin, Probiotic and L-ornithine- L Aspartate With Lactulose in Overt Hepatic Encephalopathy.
Acronym: ARGO-HEC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Qurratul Ain Jamil (Other)
Responsible Party: Sponsor-Investigator, Qurratul Ain Jamil, Assistant Professor, Department of Pharmacy Practice, Faculty of Pharmacy, The Islamia University of Bahawalpur, Islamia University of Bahawalpur
Organization: Islamia University of Bahawalpur (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 187-2023-/PHEC
Record Dates: First submitted 2025-06-09; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Overt Hepatic Encephalopathy
Keywords: Hepatic Insufficiency; Liver Cirrhosis; Rifaximin; West Haven Criteria; Grade Reversal; Lactulose; Liver Diseases
MeSH Terms: conditions — Hepatic Insufficiency; Liver Cirrhosis; Liver Diseases | interventions — Probiotics; Lactulose; Rifaximin; ornithylaspartate

STUDY DESIGN:
Intervention Model Description: A parallel study design involves assigning participants to different treatment groups, with each group receiving a distinct intervention or treatment simultaneously.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group A (Lactulose) (Active Comparator): Participant will receive lactulose syrup (120ml), 30ml (three times a day) TDS orally or by nasogastric tube (NG) for 5 days.
  Interventions: Drug: Lactulose
- Group B (Rifaximin + lactulose) (Experimental): Participant will receive Rifaximin tablet 550mg (twice daily) BID with lactulose syrup 30ml (three times a day) TDS orally or by nasogastric tube (NG) for 5 days
  Interventions: Drug: Rifaximin plus lactulose
- Group C (Probiotic + lactulose) (Experimental): Participant will receive Probiotic sachet 2g (twice daily) BID with lactulose syrup 30ml (three times a day) TDS orally or by nasogastric tube (NG) for 5 days
  Interventions: Drug: Probiotic plus lactulose
- Group D ( (L-Ornithine L- Aspartate) LOLA + Lactulose) (Experimental): Group D: LOLA (L-Ornithine L- Aspartate) concentrate for infusion (5g/10ml = 5g LOLA in 10ml clear solution) + lactulose.
  Dose: 4 ampoules (40ml) of LOLA 20g of drug diluted in 460ml of 5% dextrose was administered as an intravenous infusion at a rate of 21ml /hour (over 24 hours for 5 days) with lactulose syrup 30ml (three times a day) TDS orally or by nasogastric tube (NG)
  Interventions: Drug: L-ornithine-L-aspartate plus latulose

INTERVENTIONS:
Drug: Probiotic plus lactulose — Probiotic and lactulose will be administered per the dose and schedule specified in the arms.
  Other Names: Ecotec plus Duphalac
  Arms: Group C (Probiotic + lactulose)
Drug: Rifaximin plus lactulose — Rifaximin and lactulose will be administered per the dose and schedule specified in the arms.
  Other Names: Rifaxa plus Duphalac
  Arms: Group B (Rifaximin + lactulose)
Drug: L-ornithine-L-aspartate plus latulose — LOLA and lactulose will be administered per the dose and schedule specified in the arms.
  Other Names: Levijon concentrate for infusion plus Duphalac
  Arms: Group D ( (L-Ornithine L- Aspartate) LOLA + Lactulose)
Drug: Lactulose — Lactulose will be administered per the dose and schedule specified in the arms.
  Other Names: Duphalac
  Arms: Group A (Lactulose)

SUMMARY:
The goal of this trial is to learn if drugs in group A, B, C and D works to treat reversal of grades in people with overt hepatic encephalopathy. It will also provide information regarding safety of drugs in group A, B, C and D. The main question it aim to answer is:

Which study group is better in treating people of overt hepatic encephalopathy. Researchers will compare experimental group B (rifaximin + lactulose), group C (probiotics + lactulose) and group D (LOLA (L-Ornithine L-Aspartate) + lactulose) to control group A lactulose alone in the reversal of grades for people of hepatic encephalopathy.

Participants will:

Take drug from time of participation in the trial till the end of treatment (day 5) and grade reversal will be observed.

DETAILED DESCRIPTION:
This clinical trial aim to compare the efficacy of four groups which are group A (lactulose) as controlled group, group B (rifaximin + lactulose), group C (probiotics + lactulose)and group D (LOLA (L-Ornithine L-Aspartate) + lactulose) for treating overt hepatic encephalopathy.

Primary objective: The primary objective of our trial will be to compare the grade reversal in overt hepatic encephalopathy patients from the time of trial participation till the end of trial treatment (day 5) according to West Heaven Criteria in both control and interventional groups.

Secondary objectives:

1. To find the length of hospital stay and recovery time (in days) from hepatic encephalopathy in both control and interventional groups.
2. Monitoring of Adverse drug reactions in both control and interventional groups.
3. To assess the mortality in both control and interventional groups.

This trial is single-centered, parallel, multi-arm, 1:1:1:1 randomized, unblinded, lactulose controlled superiority clinical trial comparing the efficacy of four groups which are group A (lactulose) as controlled group, group B (rifaximin + lactulose), group C (probiotics + lactulose) and group D (LOLA (L-Ornithine L-Aspartate) + lactulose) for the treatment of overt hepatic encephalopathy.

Framework/hypothesis: The experimental group B (rifaximin + lactulose), group C (probiotics + lactulose) and group D (LOLA (L-Ornithine L-Aspartate) + lactulose) are superior to control group A lactulose alone in the reversal of grades for patients of hepatic encephalopathy.

ELIGIBILITY:
Inclusion Criteria:

1. Both male and female participants with age >18 to <80 years old at the time of consent.
2. Patients with decompensated chronic liver disease (DCLD) confirmed by ultrasound, endoscopy or blood tests associated with overt hepatic encephalopathy grade II-IV according to West Haven Criteria (WHC) will be included.
3. Patients who are unable to talk, their informed consent will be collected from first degree relative and/or legally authorized representative (LAR).
4. The subject/LAR has signed the consent/assent form authorized by the ethics committee, is willing to follow the treatment protocol, and has been informed of the purpose of the study.

Exclusion Criteria:

1. Participants with age ≤18 years old and ≥ 80 years old and those with grade1covert hepatic encephalopathy according to West Haven Criteria.
2. Patients with comorbidities including ventricular dysfunction and pulmonary edema or neurodegenerative disease (Epilepsy, Parkinson and Drug intoxication), hepatocellular carcinoma (HCC) and with major psychiatric illness (Schizophrenia).
3. Patients with presenting complaint of diarrhea will be excluded.
4. Recent or current use of sedatives or antidepressants and those who are suffering from encephalitis (viral or bacterial), Wernicke and uremic encephalopathy, stroke or brain tumor will not be included.
5. The participant is already participating in another drug trial.
6. Pregnant women will not be included.
7. Subjects suffering from terminal cancers or HIV-AIDS.
8. Participants hypersensitive to lactulose, rifaximin, LOLA and probiotics or any of its excipients will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-04-21 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Number of participants of overt hepatic encephalopathy are treated by observing reversal in grades by using West Haven Criteria. | From the time of enrollment till the end of treatment (day 5) in the trial.
  To compare the efficacy of group B (rifaximin + lactulose), group C (probiotics + lactulose) and group D (LOLA (L-Ornithine L-Aspartate) + lactulose) with group A (lactulose) as controlled group for the treatment of overt hepatic encephalopathy, grade reversal is examined from the time of participation in the trial till the end of treatment (day 5) according to West Heaven Criteria.
  The West Haven criteria are a widely used system for classifying the severity of hepatic encephalopathy. It grades the condition from Grade 0 (minimal or no symptoms) to Grade 4 (coma) based on the patient's level of consciousness, intellectual function, and behavior.

SECONDARY OUTCOMES:
Time of recovery from encephalopathy (Days) | Time of participation in the study assessed up to 5 days.
  Time of recovery from encephalopathy is defined as the time taken (in days) to recover from grade 2 or above mental state grade to grade 1 or below.
Liver disease severity | time of participation in the trial till the end of treatment (day 5)
  Severity of liver disease will be evaluated by Child-pug class. The Child-Pugh score is a clinical tool designed to evaluate the severity of chronic liver disease, including conditions like hepatic encephalopathy (HE). It classifies patients into three categories: A, B, and C, reflecting the degree of liver dysfunction. A higher score corresponds to more severe liver disease and a worse prognosis. This scoring system aids in assessing liver damage, predicting patient survival, and informing treatment options, such as the necessity for liver transplantation.
  Interpretation:
  Child-Pugh Class A: 5-6 points, indicating well-compensated liver disease. Child-Pugh Class B: 7-9 points, indicating moderately impaired liver function. Child-Pugh Class C: 10-15 points, indicating severely compromised liver function and decompensation.
length of hospital days | time of participation in the study till the patient is discharged or died or till 28 days whichever occur earlier.
  To find length of in- hospital stay (days) is defined as the time patient spent in hospital setting until he/she is discharged.

CONTACTS AND LOCATIONS:
Overall Officials: QurratulAin Jamil, PhD, Principal Investigator — The Islami University of Bahawalpur
Locations (1):
- Bahawal Victoria Hospital, Bahawalpur, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shahbaz A, Jamil Q, Iqbal SM, Jamil MN, Khan JA, Aufy M. Comparison of efficacy of rifaximin, probiotics and L-ornithine L-aspartate in overt hepatic encephalopathy: a randomized, phase IV, lactulose controlled clinical trial. Trials. 2025 Nov 21;26(1):534. doi: 10.1186/s13063-025-09173-2. PMID 41272855

DOCUMENTS (1):
  • Informed Consent Form (2023-08-25): https://cdn.clinicaltrials.gov/large-docs/94/NCT07037394/ICF_000.pdf